CLINICAL TRIAL: NCT04869917
Title: Behavioral Nudges for Diabetes Prevention (BEGIN) Trial in Primary Care
Acronym: BEGIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Matthew J O'Brien, Associate Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00212461
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: This study will utilize a 2x2 factorial design to test the effectiveness of the two proposed interventions on outcomes. Each of the participating clinical sites will be randomized to one of 4 treatment conditions. Employing a full factorial design, the participating clinics sites will be randomized to 1 of the following 4 treatment conditions: a) prediabetes decision aid intervention alone; b) text messaging intervention alone; c) both interventions; and d) usual care [i.e. neither intervention].
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Decision Aid intervention (Experimental): Health Educators (HEs) will meet briefly with eligible participants after each office visit to review a prediabetes decision aid which reviews information about the benefits and risks of intensive lifestyle intervention and metformin.
  Interventions: Behavioral: Decision Aid intervention
- Text Messaging intervention (Experimental): Participants will receive biweekly messages throughout the 12-month trial. Automated messages will be sent using an existing secure text messaging platform.
  Interventions: Behavioral: Text Messaging intervention
- Decision Aid intervention + Text Messaging intervention (Experimental): Health Educators (HEs) will meet briefly with eligible participants after each office visit to review a prediabetes decision aid. Additionally, participants will receive biweekly messages throughout the 12-month trial. Automated messages will be sent using an existing secure text messaging platform.
  Interventions: Behavioral: Decision Aid intervention; Behavioral: Text Messaging intervention
- Usual Care (Placebo Comparator): Usual care includes no additional intervention above the care routinely provided at the clinical partner site, Erie Family Health Center.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Decision Aid intervention — * Displays information about the benefits and risks of ILI and metformin
  * Asks open-ended questions: "What am I willing to do to prevent T2D?" and "What do I need to prevent T2D?"
  * Prompts patients to commit to immediate next steps
  * Health educator schedules interested patients for first ILI session or sends message to provider about patients' interest in starting metformin, if chosen
  Arms: Decision Aid intervention; Decision Aid intervention + Text Messaging intervention
Behavioral: Text Messaging intervention — * Defines prediabetes and includes individualized A1c values
  * Present benefits and risks of intensive lifestyle intervention and metformin
  * States that other prediabetic Erie patients are adopting intensive lifestyle intervention and metformin
  * Encourages initiating intensive lifestyle intervention or discussing metformin with provider
  * Include selected behavioral content from diabetes prevention program
  * Initial message with automatic opt-in, allows opt-out for messages
  * Subsequent messages include: information about T2D risk and treatments; prompts to directly schedule intensive lifestyle intervention or office visit to discuss metformin; selected behavioral content from diabetes prevention programming
  Arms: Decision Aid intervention + Text Messaging intervention; Text Messaging intervention
Behavioral: Usual Care — Patients receiving care at non-intervention clinic sites will not be exposed to treatment intervention.
  Arms: Usual Care

SUMMARY:
A large body of research has demonstrated that intensive lifestyle interventions and metformin are effective treatments to prevent or delay diabetes among high-risk adults, yet neither treatment is routinely used in practice. The Behavioral Nudges for Diabetes Prevention (BEGIN) Trial will test two low-touch interventions designed to motivate adoption of these treatments to prevent diabetes. Given that 38% of U.S. adults have prediabetes, the proposed study has potential for large public health impact by testing pragmatic, scalable, and sustainable approaches based in primary care to promote evidence-based treatment for this common condition.

DETAILED DESCRIPTION:
Large randomized trials have found that intensive lifestyle interventions (ILI) and metformin are safe and effective treatment options for promoting modest weight loss and preventing type 2 diabetes (T2D) among adults with prediabetes. However, these treatments are rarely used in practice, and little existing research has focused on patient-centered approaches for promoting their use. One potential approach, behavioral nudges, involves manipulating health messages and treatment options to make behavior change more likely and easier to enact. While a large body of evidence suggests that behavioral nudges are effective, they have not been definitively studied for T2D prevention. The study team will address this critical knowledge gap by conducting the Behavioral Nudges for Diabetes Prevention (BEGIN) Trial. The proposed study will take place in primary care clinics, whose unprecedented reach and regular interaction with prediabetic adults make this an ideal setting for translational T2D prevention research. This definitive study will test two low-touch interventions: 1) prediabetes decision aid intervention consisting of a prediabetes decision aid designed to nudge uptake of evidence-based treatments and delivered by health educators; and 2) text messaging intervention consisting of text messages that deliver similar information and use the same behavioral nudges. The proposed R18 study will accomplish the following specific aims to determine the most effective low-touch intervention that promotes maximal treatment adoption and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18-80 years)
* with prediabetes
* overweight/obesity (BMI ≥25kg/m2)
* patients who speak English or Spanish

Exclusion Criteria:

* type 2 diabetes
* dementia
* serum creatinine >1.4mg/dL in women and >1.5mg/dL in men
* current use of oral corticosteroids
* current pregnancy
* uncontrolled hypertension (≥180/100mmHg)
* history of metformin use
* no office visits during the last 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 months
  Mean differences in weight (lbs) between treatment arms will be evaluated using mixed models adjusted for clinic site, time between visits, sex, age, race/ethnicity, and baseline cardiometabolic markers

SECONDARY OUTCOMES:
Participant initiation of treatment to intensive lifestyle (ILI) or Metformin | 12 months
  The number of participants that initiate ILI, Metformin, or both treatments at follow-up which will be assessed in the following ways. Because initiation of metformin requires a provider prescription, this will be assessed pragmatically using the electronic health record (EHR) and confirmed by participant self-report of taking at least 1 dose. Attendance logs will be used to confirm whether participants attended at least 1 ILI session. Those who received a prescription for metformin but do not take any doses will not be considered to have initiated treatment. Similarly, those who are referred to ILI but do not attend any sessions will not be classified as initiating treatment. Receiving a provider's prescription for metformin or referral for ILI without initiating treatment will be an exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, MD, Principal Investigator — Associate Professor
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vargas MC, Pineda GJ, Talamantes V, Toledo MJL, Owen A, Carcamo P, Gibbert W, Ackermann RT, Kandula NR, Cameron KA, Siddique J, Williams GC, O'Brien MJ. Design and rationale of behavioral nudges for diabetes prevention (BEGIN): A pragmatic, cluster randomized trial of text messaging and a decision aid intervention for primary care patients with prediabetes. Contemp Clin Trials. 2023 Jul;130:107216. doi: 10.1016/j.cct.2023.107216. Epub 2023 May 9. PMID 37169219